CLINICAL TRIAL: NCT02758028
Title: Helping Youth Smokers Stop Smoking Through the Youth Quitline Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: YouthQuitline
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
Keywords: Youth; Adventure-based training; WhatsApp messages
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief counseling (Other): Peer counselling is delivered based on the queries and the needs of individual clients, according to the smoking status, dependency level and the perceived barriers of each individual with the use of motivational intervention approach. Counsellors will emphasizes the identification, use, and modification of personally relevant coping strategies. Advice will be provided on overcoming expected difficulty, withdrawal symptoms and relapse prevention during quitting.
  The subjects will be followed up at 1-week, 1-, 3-, 6-, 9-, 12- and 24-month via telephone assessing their smoking status and reinforce intervention.
  Interventions: Behavioral: Brief counseling

INTERVENTIONS:
Behavioral: Brief counseling — Peer counselling is delivered based on the queries and the needs of individual clients, according to the smoking status, dependency level and the perceived barriers of each individual with the use of motivational intervention approach.
  The subjects will be followed up at 1-week, 1-, 3-, 6-, 9-, 12- and 24-month via telephone assessing their smoking status and reinforce intervention.

SUMMARY:
The aims of the present study are:

1. To raise the awareness of smoking cessation service among youth smokers in Hong Kong;
2. To provide smoking cessation quitline service to youth smokers; and
3. To provide training to teenagers as peer smoking cessation counsellors.
4. To examine the effectiveness of adventure-based training and WhatsApp messages in helping youth smokers to quit

DETAILED DESCRIPTION:
In Hong Kong, the demand of smoking cessation service of Youth was increasing in the past 10 years, the first youth-oriented smoking cessation hotline "Youth Quitline" was established in 2005. From August 2005 to July 2016, "Youth Quitline" has received over 9,267 telephone inquiries and provided telephone smoking cessation counselling for 1,952 youth smokers.

Youth smokers are recruited using the reactive and proactive strategies. The operation hours of Quitline service are weekdays from 17:00 to 21:00 and on weekends from 14:00 to 20:00. A questionnaire asking the smoking status, reason of smoking, dependency level, knowledge, attitude and practice of smoking or quitting at baseline, the perceived barriers of the smokers and the use of other tobacco products were designed to assess the status of participants, brief counselling with the use of motivational intervention approach is delivered during the phone call.

Telephone counseling at 1-week, 1-month, 3-month, 6-month, 9-month, 12-month and follow-up at 24-month are conducted with the participants to assess their smoking status (by questionnaire) and reinforce intervention (encourage quitting and providing quitting tips). Self-reported quitters who have quitted smoking for at least 7 days at 6-month are invited to perform saliva cotinine test (using NicAlert strip) plus exhaled carbon monoxide text to validate the smoking status.

A qualitative interview will be conducted to investigate the use of other tobacco products of the Youth Quitline participants, and aimed to find out their smoking patterns and feelings of using these products, and how these products might affect quitting or smoking, and how the protest activates influence the smoking behaviors among the youth smokers.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 25 or below
* Able to communicate in Chinese (Cantonese)
* Smoked in the past 30 days

Exclusion Criteria:

* Have difficulty to communicate via telephone
* Having queries irrelevant to tobacco control

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-08; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
7-days point prevalence smoking abstinence at 6-month | 6-month follow-up
  7-days point prevalence smoking abstinence is measured at 6-month. A questionnaire asking smoking status, quitting experience and difficulty in quitting was designed to assess the self-reported smoking abstinence at 6-month.

SECONDARY OUTCOMES:
Bio-chemical validated smoking abstinence at 6-month | 6-month follow-up
  Bio-chemical validated smoking abstinence is measured at 6-month. The participants who claim to have quitted smoking for at least 7 days are invited for biochemical validation (measurement of saliva cotinine level and exhaled carbon monoxide level) at 6-month. The participants are need to get the results of CO≤ 4ppm, and continine level ≤30 ng/ml as passing results.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)